CLINICAL TRIAL: NCT07374315
Title: A Family-based Intervention Approach to Address Weight Gain in Pediatric Leukemia Survivors
Brief Title: Weight Gain in Pediatric Leukemia Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202512147
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Pediatric Acute Lymphoblastic Leukemia; Pediatric Acute Lymphoblastic Leukemia in Remission; Pediatric Obesity
Keywords: Leukemia; Lymphoblastic Leukemia; Weight Management; Late Effects; Health Behaviors; Healthy Habits
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pediatric Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Forty patient-caregiver dyads (total of 80 participants) will be enrolled and randomized 1:1 to Arm A or Arm B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Educational Resources (Active Comparator): Participants will be provided direction to NIH educational resources over the course of the intervention. Both programs provide resources to improve nutrition, increase physical activity, limit screen time, and improve sleep and consist of online, free, assessable educational materials. Patients and caregivers will be reminded of this resource at their monthly clinic appointments for 6 months after their first study visit.
  Interventions: Behavioral: NIH Educational Resources; Behavioral: FitBit Ace; Behavioral: WashU Extended Learning Canvas
- Arm B: Modified Guided Self-Help Family Intervention (mL-GSH) (Experimental): Participants will complete the Modified Guided Self-Help Family Intervention for survivors of leukemia (mL-GSH). ML-GSH is a six-session intervention to be delivered during appointments. Patients will have 6 months to complete the curriculum (may be up to 9 months to account for scheduling concerns).
  Interventions: Behavioral: Modified Guided Self-Help Family Intervention; Behavioral: FitBit Ace; Behavioral: WashU Extended Learning Canvas

INTERVENTIONS:
Behavioral: Modified Guided Self-Help Family Intervention — Patients and their caregivers will be led through mL-GSH in six sessions over the course of 6-9 months. Content is informed by priorities of caregivers and survivors of pediatric leukemia. The curriculum relies on participants identifying habits to monitor independently and supplementing their engagement with additional materials.
  Other Names: mL-GSH
  Arms: Arm B: Modified Guided Self-Help Family Intervention (mL-GSH)
Behavioral: NIH Educational Resources — Patients and their caregivers will be provided education materials from the NIH. The educational resources are We Can! a National Institute of Health educational resource designed for parents, caregivers, and communities to help children ages 8 through 13 improve their health and Take Charge of Your Health which is designed to provide education to teenagers to improve their health
  Arms: Arm A: Educational Resources
Behavioral: FitBit Ace — Patients will be provided with a FitBit Ace. FitBit Ace will be worn by patients to track physical activity.
Behavioral: WashU Extended Learning Canvas — All caregivers will be provided access to WashU Extended Learning Canvas. The WashU Extended Learning Canvas will have an online support group for caregivers to engage in with other caregivers in the trial.

SUMMARY:
This is a trial assessing the efficacy of two weight maintenance programs for children with acute lymphoblastic leukemia (ALL) and the patients' caregivers. Patients and their caregivers will be randomized 1:1 to Arm A, a non-intensive educational intervention using National Institute of Health (NIH) Educational Resources (We Can! for children 8-13 and Take Charge of Your Health for teenagers 14-18), or Arm B, a Modified Guided Self-Help Family Intervention for Leukemia patients (mL-GSH). Outcomes will be assessed through activity trackers, obesity biometrics, and nutrition and physical activity assessments.

ELIGIBILITY:
Patient Eligibility Criteria:

* Must have a diagnosis of ALL (T or B cell).
* Must be receiving standard of care maintenance chemotherapy or be within 6 months of having concluded maintenance chemotherapy at the time of enrollment.
* Must be at least 6 years of age and no older than 18 years of age at time of enrollment.
* Must be able to speak and understand English.
* Must have a caregiver who is participating in this study.
* Must be able to perform some level of exercise (e.g., a brisk walk for at least five minutes) as determined by self-report.
* Must not have severe developmental delay/intellectual disabilities (such as Trisomy32, severe presentations of autism spectrum disorder) or significant mental illness (such as active suicidal ideation, psychotic symptoms, manic or hypomanic episodes, or severe substance use disorder) that may interfere with ability to participate in modified Family Based Therapy (FBT).
* Patients 10 and older must have a negative SCOFF screen for disordered eating (Score of 2 or more would disqualify the patient and require discussion with primary team)
* Must be able to understand and willing to sign an IRB-approved written informed consent document or be able to provide verbal assent along with written consent provided by a legally authorized representative.

Caregiver Eligibility Criteria:

* Self-reported as the primary caregiver of a pediatric patient diagnosed with ALL who is also participating in this study.
* Must be at least 18 years of age.
* Must be able to speak and understand English.
* Must be able to perform some level of exercise (e.g., a brisk walk for at least five minutes) as determined by self-report
* Must be able to understand willing to sign an Institutional Review Board (IRB)-approved written informed consent document.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight Z score | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Participant's weight Z score is a statistical value that indicates how the participant's weight for their age and sex compares to the average weight for that population which is obtained from Center for Disease Control (CDC) growth Charts
Changes in weight Z score | From start of study through end of study (estimated total time frame 12-15 months)
  Participant's weight Z score is a statistical value that indicates how the participant's weight for their age and sex compares to the average weight for that population which is obtained from CDC growth Charts. Changes in weight Z score from start to end of the study will be analyzed by changes in summary statistics (mean, median, and standard deviation) across timepoints.
BMI Z Score | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Participant's BMI Z score is a statistical value that indicates how the participant's BMI for their age and sex compares to the average BMI for that population which is obtained from CDC growth Charts
Changes in BMI Z Score | From start of study through end of study (estimated total time frame 12-15 months)
  Participant's BMI Z score is a statistical value that indicates how the participant's BMI for their age and sex compares to the average BMI for that population which is obtained from CDC growth Charts. Changes in BMI Z score from start to end of the study will be analyzed by changes summary statistics (mean, median, and standard deviation) across timepoints.
Changes in Cholesterol | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Changes in cholesterol (total, LDL, and HDL levels) will be analyzed via summary statistics (means, medians, and standard deviation) at each of the endpoints.
Changes in HbA1c | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Changes in HbA1c will be analyzed via summary statistics (means, medians, and standard deviation) at each of the endpoints.
Changes in Albumin | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Changes in albumin will be analyzed via summary statistics (means, medians, and standard deviation) at each of the endpoints.

SECONDARY OUTCOMES:
Changes in activity intensity assessed by Fitbit Ace Smartwatch using the Freedson age-adjusted equation | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  The Freedson age-adjusted equation is used to estimate maximum heart rate based on age and then is used to classify activity intensity by the heart rate of the activity.
Changes in activity levels as measured by PAQ-C assessments | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Activity levels will be assessed by participants' changes in scores across different timepoints on Physical Activity Questionnaire for Older Children (PAQ-C). The PAQ-C is a self-administered, 7 day recall questionnaire designed to assess physical activity of children by proving a summary score of moderate to vigorous physical activity (MVPA). The mean PAQ-C score is interpreted as follows: 1.0-1.9 low physical activity, 2.0-2.9 moderate-low activity, 3.0-3.9 moderate activity, and 4.0-5.0 high activity. A higher score indicates a higher activity level.
Changes in activity levels as measured by PAQ-A assessments | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Activity levels will be assessed by participants' changes in scores across different timepoints on Physical Activity Questionnaire for Adolescents (PAQ-A). The PAQ-A is a self-administered, 7 day recall questionnaire designed to assess physical activity of adolescents by proving a summary score of moderate to vigorous physical activity (MVPA). The mean PAQ-A score is interpreted as follows: 1.0-1.9 low physical activity, 2.0-2.9 moderate-low activity, 3.0-3.9 moderate activity, and 4.0-5.0 high activity. A higher score indicates a higher activity level.
Changes in health behaviors as measured by the Health Behaviors Survey | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  The health behaviors survey assesses average daily activity level, screen time, sweetened beverage consumption, and fruit and vegetables consumption to determine if patients are compliant with American Academy of Pediatrics Recommendation. 44% of childhood cancer survivors are active more than 60 minutes a day, 40% engage in less than 1 hour of screen time, 34% consume sweetened beverages and 4% consume more than one serving of fruits and vegetables.
Changes in 24-hour dietary recall as measured by ASA24 | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention. Estimated total time frame of 12-15 months.
  Patient and caregiver feeding habits will be assessed by their responses to a 24 hour dietary recall through the Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). ASA24 is a web-based, automated dietary recall tool that uses images and prompts. The ASA24 produces automated nutrient and food group data on participant's diet, a Respondent Nutrition Report (RNR). The RNR data will be used to generate a Healthy Eating Index score ranging from 0-100 with higher scores indicating closer alignment to the Dietary Guidelines for Americans. Between group differences between Arm A and Arm B will be compared via various statistical methods.
Changes in health behaviors as measured by Childhood Feeding Questionnaire | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Changes in health behaviors will be assessed by caregivers' responses to the Child Feeding Questionnaire (CFQ and CFQ-teen) across different timepoints. The Child Feeding Questionnaire is a 31-item questionnaire using a 5-point Likert scale to assesses parents/caregivers' beliefs, attitudes, and practices surrounding feeding and their perceptions of their child's weight and eating behavior. The CFQ includes seven subscales. Subscales are scored from 1-5 with general guidelines for interpreting subscale scores as follows: 1.0-1.9 very low use of that feeding practice/low perception, 2.0-2.9 below average/mild expression, 3.0-3.9 moderate/typical parental level, and 4.0-5.0 high use or strong perception/belief.
Changes in Health Habits Survey | Enrollment, during intervention (4 months after enrollment), end of intervention (6 months after enrollment (may be up to 9 months)), and 6 months after end of intervention (estimated total time frame of 12-15 months)
  Changes in answers to the Health Habits Survey will be assessed by caregivers and patients' responses to the survey at different timepoints. The Health Habits Survey is an assessment consisting of four questions evaluating health behaviors using 4-point Likert scales. These behaviors include daily activity level (not very often, <30 min a day, 30-60 min a day, and ≥ 60 min a day), screen time ( ≥2 hr a day, 1-2 hr a day, 30-60 min a day, and not very often), sweetened beverage consumption ( ≥3 a day, two a day, one a day, and not very often), and fruit and vegetable consumption (0-1, 1-2, 3-4, or >4 times a day.). The investigators will consider percentage of children whose health habits align with American Academy of Pediatric recommendations - 5 fruits and vegetables per day, 2 hours or less of screen time, 1 hour of physical activity, 0 sweetened beverages consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Ferris, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be deidentified and accessible following publication of study results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after publication of study results with no end date for data sharing.
Access Criteria: Data will be shared with any individual who wishes to have access to the data for any purpose. Data will be included in supplementary materials of publication. Data will also be available by request to the corresponding authors of the publication.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu